CLINICAL TRIAL: NCT06905704
Title: Retrospective-prospective Observational Monocentric Study Evaluating the Impact of Stem Cell Donation on Unrelated and Related Donors' Health.
Brief Title: Impact of Stem Cell Donation on Unrelated and Related Donors' Health.
Acronym: HPCDON
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Claudia Del Fante, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: HPCDON
Record Dates: First submitted 2025-03-21; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-02

CONDITIONS: Stem Cell Donors
Keywords: stem cell donors, safety, transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Haematopoietic stem cell donation represents a unique chance for curing patients affected with onchohaematologic and inherited diseases.If a related donor is unavailable a unrelated donor must be used. For both categories an accurate physical and laboratory examination is mandatory to establish the eligibility to bone marrow or peripheral blood stem cell collection since side effects related to donation may occur. To ensure high standards of safety and satisfaction of unrelated stem cells donors dedicated guidelines are available. On the other hand, there is no unambiguous guidance on the management of the related donor and published data on donation and long term follow-up are scarce.

DETAILED DESCRIPTION:
The study, for the retrospective part, aims to report the experience in family and registry donor management at Transfusion Service from 2016 to 2022 (enrollment, stem cell donation, 30-day follow-up) and, for the prospective part, to continue monitoring on donors who will be enrolled in the next five years (2023 to 2028).

ELIGIBILITY:
Inclusion Criteria:

* Family donors ≥18 years referred by the Hematology and Oncohematology Transplant Center Pediatric of the Foundation of Centro Donatori -SIMT, following the national and international guidelines after medical evaluation
* Volunteer donors from IBMDR registry ≥18 years, following the national and international guidelines after medical evaluation

Exclusion Criteria:

* Donors 18 < years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: stem cell donors
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
safety of stem cell donation | From enrollment to 30 days after stem cell donation
  The proportion of overall serious adverse reactions/events (number of patient-reactions out of the total number of patients)

SECONDARY OUTCOMES:
peripheral stem cells analysis | From enrollment to 30 days after stem cell donation
  Measurement of blood counts and CD34+ cells pre-donation and in the collected product
lymphocyte analysis | From enrollment to 30 days after stem cell donation
  Cytofluorimetric analysis of lymphocyte subpopulations (CD4, CD8, CD4/8 ratio) at donor enrollment
CBC analysis | From enrollment to 30 days after stem cell donation
  CBC examination at different measurement times

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy